CLINICAL TRIAL: NCT05359432
Title: Comparison of Empaglifozin and Vildagliptin in Efficacy and Safety in Type 2 Diabetes Mellitus
Brief Title: Comparison of Empaglifozin and Vildagliptin in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Responsible Party: Principal Investigator, Jaffer Bin Baqar, Dr. Asima Niazi, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK_01
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes Mellitus; Empagliflozin; Vildagliptin; Efficacy; Safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Vildagliptin (Experimental)
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Empagliflozin — Receiving allocated drug dosage as per clinical needs
  Arms: Empagliflozin
Drug: Vildagliptin — Receiving allocated drug dosage as per clinical needs
  Arms: Vildagliptin

SUMMARY:
The aim of this study is to perform a comparison of the efficacy and safety of empagliflozin and vildagliptin in patients with Type 2 Diabetes Mellitus

open labelled, multi-centric, parallel, randomized control trial

In Type 2 Diabetes patients, impact of empagliflozin (10 mg once or twice daily) versus vildagliptin (50 mg once or twice daily) assessed for Efficacy & safety parameters to be measured at both the baseline and 24-week visits.

DETAILED DESCRIPTION:
Background:

Diabetes is a rampant disease that keeps on getting more and more people affected each year. Over 200 million people have been affected worldwide due to this disorder, and many have contracted various cardiovascular complications due to uncontrolled diabetes. Though an easily manageable disease, if left untreated, diabetes can be fatal. Therefore, it is necessary to have drugs available which control diabetes and also limit the progression of complications that could arise due to it.

Objective:

The aim of this study is to perform a comparison of the efficacy and safety of empagliflozin and vildagliptin in patients with Type 2 Diabetes Mellitus

Methods:

open labelled, multi-centric, parallel, randomized control trial to be conducted at the Department of Diabetes & Endocrinology of two tertiary care hospitals in Karachi, Pakistan.

The Participants will undergo screening and then were randomized into two groups. The first group received empagliflozin (10 mg once or twice daily), and the second group received vildagliptin (50 mg once or twice daily. HbA1c, High-density lipoprotein (HDL) levels., Systolic blood pressure, fasting blood glucose, and body weight will be measured at both the baseline and 24-week visits.

ELIGIBILITY:
Inclusion Criteria:

Female and Male Patients of age 30-65 years with confirmed diagnosis of "type 2 diabetes mellitus".

Uncontrolled type 2 diabetes mellitus (> 7% HbA1c patients on monotherapy of metformin for the past three months on a fixed dose of 1500 mg /day along with lifestyle modifications were included in this study.

BMI ranges from 18-45 kg/m2 were considered fit for this study. eGFR ≥ 60 ml/min/1.73 m2

Exclusion Criteria:

Pregnant female or female patients planning to conceive during the study period were excluded from this study.

"Type 1 diabetes" or "secondary diabetes" resulting from specific causes Patients with advanced diabetic complications. Patients with any other terminal disease(s) requiring long-term medications. Patients involved in other trials on therapy with SGLT-2i or DPP4-I 3 months before study enrollment Patients on insulin or any other oral hypoglycemic drugs except metformin. Serum creatinine levels ≥ 1.3 mg/dl in women and ≥ 1.4 mg/dl in men

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin A1c (HbA1c) | 24 weeks
High-density lipoprotein (HDL) levels | 24 weeks
Systolic blood pressure | 24 weeks
Fasting blood sugars | 24 weeks
Bodyweight | 24 weeks
Serum creatinine | 24 weeks
Serum glutamic-pyruvic transaminase (SGPT) | 24 weeks
Low-density lipoprotein cholesterol | 24 weeks
Total cholesterols | 24 weeks
Serum triglycerides | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Diabetes and Endocrinology at Sindh Government Hospital New Karachi & Dr. Riasat Medical Center Allah Wala Town, Karachi, Pakistan, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Study data with CRF
Supporting Information: Study Protocol, ICF
Time Frame: In 1 month for 1 year

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Deshpande AD, Harris-Hayes M, Schootman M. Epidemiology of diabetes and diabetes-related complications. Phys Ther. 2008 Nov;88(11):1254-64. doi: 10.2522/ptj.20080020. Epub 2008 Sep 18. PMID 18801858
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2005 Jan;28 Suppl 1:S37-42. doi: 10.2337/diacare.28.suppl_1.s37. No abstract available. PMID 15618111
- [Background] Strodl E, Kenardy J. Psychosocial and non-psychosocial risk factors for the new diagnosis of diabetes in elderly women. Diabetes Res Clin Pract. 2006 Oct;74(1):57-65. doi: 10.1016/j.diabres.2006.02.011. Epub 2006 Apr 11. PMID 16584801
- [Background] Lin YK, Gao B, Liu L, Ang L, Mizokami-Stout K, Pop-Busui R, Zhang L. The Prevalence of Diabetic Microvascular Complications in China and the USA. Curr Diab Rep. 2021 Apr 9;21(6):16. doi: 10.1007/s11892-021-01387-3. PMID 33835284